CLINICAL TRIAL: NCT05903547
Title: Glue Versus Subcuticular Suture for Cesarean Closure: a Randomized Control Trial
Brief Title: A Skin Glue Versus Subcuticular Suture for Cesarean Closure Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Russell Miller, Sloane Hospital for Women Associate Professor of Prenatal Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAT9584
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Section; Complication; Wound
Keywords: Complications; Wound; Hematoma; Surgical Incision
MeSH Terms: conditions — Wounds and Injuries; Hematoma; Surgical Wound | interventions — Sutures

STUDY DESIGN:
Intervention Model Description: Women undergoing cesarean delivery will be recruited and randomized to skin closure with either the Dermabond Prineo system or standard subcuticular suture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Dermabond Prineo Group (Active Comparator): At time of cesarean delivery, patients in the Dermabond Prineo group will undergo skin closure with the Dermabond Prineo skin adhesive system.
  Interventions: Device: Dermabond Prineo
- Suture Group (Placebo Comparator): At time of cesarean delivery, patients in the Suture group will undergo skin closure with standard subcuticular suture.
  Interventions: Other: Suture

INTERVENTIONS:
Device: Dermabond Prineo — For subjects in the Dermabond Prineo group, the Dermabond Prineo system will be applied to the skin for skin closure under manufacturer's guidelines.
  Arms: Dermabond Prineo Group
Other: Suture — For subjects in the Suture group, the skin will be closed with the standard subcuticular suture method.
  Arms: Suture Group

SUMMARY:
The aim of this study is to compare cesarean incision outcomes between patients with incision closed with the Dermabond Prineo system compared to standard subcuticular suture.

DETAILED DESCRIPTION:
The purpose of this study is to assess patient satisfaction with their incision after undergoing cesarean delivery. Patient satisfaction with their cesarean scar at 4-6 weeks after their surgery will be compared amongst women receiving skin closure with the Dermabond Prineo skin adhesive system versus standard subcuticular suture. Dermabond Prineo has been shown to have improved cosmesis outcomes in non-obstetric populations but has not yet been studied for women receiving cesarean section. In addition to scar appearance, outcomes such as wound infection, postoperative pain, and operative time will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years or older
* All women scheduled for primary or repeat cesarean deliveries
* All women undergoing intrapartum or antepartum cesarean delivery
* Pfannenstiel skin incision
* Birth of a live infant at time of cesarean delivery

Exclusion Criteria:

* Vertical skin incision
* Cesarean hysterectomy
* Emergency or stat cesarean delivery excluding standard preoperative preparation measures (i.e., use of Chlorhexidine skin prep, vaginal prep, etc)
* Intrapartum stillbirth
* Planned postpartum follow up at another facility
* Contraindications to routine postpartum pain medications
* Adhesive or tape allergy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell Miller, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center/NYP, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Goto S, Sakamoto T, Ganeko R, Hida K, Furukawa TA, Sakai Y. Subcuticular sutures for skin closure in non-obstetric surgery. Cochrane Database Syst Rev. 2020 Apr 9;4(4):CD012124. doi: 10.1002/14651858.CD012124.pub2. PMID 32271475
- [Background] Dumville JC, Coulthard P, Worthington HV, Riley P, Patel N, Darcey J, Esposito M, van der Elst M, van Waes OJ. Tissue adhesives for closure of surgical incisions. Cochrane Database Syst Rev. 2014 Nov 28;2014(11):CD004287. doi: 10.1002/14651858.CD004287.pub4. PMID 25431843
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Fleisher J, Khalifeh A, Pettker C, Berghella V, Dabbish N, Mackeen AD. Patient satisfaction and cosmetic outcome in a randomized study of cesarean skin closure. J Matern Fetal Neonatal Med. 2019 Nov;32(22):3830-3835. doi: 10.1080/14767058.2018.1474870. Epub 2018 May 24. PMID 29739243
- See also: Dermabond Prineo — https://www.jnjmedtech.com/sites/default/files/user_uploaded_assets/pdf_assets/2020-10/DERMABOND%C2%AE%20PRINEO%C2%AE%20Skin%20Closure%20System%20Brochure%20113568-190506.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dermabond Prineo Group | Suture Group
Started | 73 | 78
Completed | 73 | 78
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dermabond Prineo Group | Suture Group | Total
Number analyzed (Participants) | 73 | 78 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (5.3) | 33.1 (5.6) | 34 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 78 | 151
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 42 | 83
  Not Hispanic or Latino | 27 | 33 | 60
  Unknown or Not Reported | 5 | 3 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 17 | 29
  White | 25 | 25 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 33 | 35 | 68
Region of Enrollment [Number; unit: participants]
  United States | 73 | 78 | 151

OUTCOME MEASURES:

1. Primary Outcome: Patient Scar Satisfaction Scale Score
Description: The patient's satisfaction with their cesarean incision will be assessed using the validated Patient Scar Assessment Scale (PSAS) questionnaire. The PSAS is a 6-item questionnaire that is scored on a 1 (no complaints/as normal skin) to 10 (worst imaginable/very different from normal skin) scale. Total scores range from 6-60, with a lower score indicating a greater level of patient satisfaction.
Time Frame: Assessed at 6-weeks postpartum
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Dermabond Prineo Group | Suture Group
Number analyzed (Participants) | 73 | 78
score on a scale | 13 [9 to 20] | 13.5 [9 to 21.8]

2. Secondary Outcome: Incidence of Surgical Site Infection (SSI)
Description: A composite of surgical site infection (SSI) will be assessed. This composite will include superficial and deep SSI, endometritis, wound separation from any cause, and/or fascial dehiscence.
Time Frame: Up to 6 weeks post-surgery
Reporting Status: Not Posted

3. Secondary Outcome: Skin Closure Time
Description: The skin closure time will be assessed.
Time Frame: Intraoperative
Reporting Status: Not Posted

4. Secondary Outcome: Operative Time
Description: The total operative time will be assessed.
Time Frame: Intraoperative
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 weeks post-surgery
Arm/Group | Dermabond Prineo Group | Suture Group
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/78
Serious Adverse Events (participants affected / at risk) | 5/73 | 11/78
Other Adverse Events (participants affected / at risk) | 9/73 | 8/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dermabond Prineo Group (N=73) | Suture Group (N=78)
Prolonged Hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Readmission or presentation to ED (Pregnancy, puerperium and perinatal conditions) | 5 | 9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dermabond Prineo Group (N=73) | Suture Group (N=78)
Surgical site complication (Surgical and medical procedures) | 9 | 8 — Surgical site infection or complication for delivery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/47/NCT05903547/Prot_SAP_001.pdf